CLINICAL TRIAL: NCT05084950
Title: Informing the Population of Their Level of Protection Against COVID-19 in Monaco: a Prospective Study (MonaVacc)
Acronym: MonaVacc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Scientifique de Monaco (Other)
Collaborators: Department of Health Affairs, Monaco (Unknown)
Responsible Party: Sponsor
Other Study IDs: PRO_CSM_02_2021
Record Dates: First submitted 2021-10-19; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV-2; COVID-19; Vaccines; Antibody
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vaccines against the coronavirus type 2 causing severe acute respiratory syndrome Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) have been created in a short period of time due to the rapid spread of the virus. These vaccines use different and sometimes innovative technologies, such as the use of ribonucleic acid (RNA), or a non-replicating viral vector. Efficacy ranging from 70-90% in the first weeks after the second injection of these vaccines has been reported, with side effects whose causality remains to be determined.

DETAILED DESCRIPTION:
Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)

ELIGIBILITY:
Inclusion Criteria:

* Participant must live in the Principality of Monaco
* Deliver a written consent to participate to the study
* And/Or Have been infected with SARS-CoV-2
* And/Or Have been, or are about to be, vaccinated against SARS-CoV-2

Exclusion Criteria:

- None of the above

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a single-centre prospective observational study in the general population of the Principality of Monaco, attending the community public health center of Monaco, for Covid testing and/or vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Covid-19 Neutralizing Antibodies Measurment | 24-month period
  Inform any individual who has been infected with or vaccinated against Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) have about their level of immune protection, through a bi-annual follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Centre National de Depistage - Espace Leo Ferre, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: Undecided